CLINICAL TRIAL: NCT00547053
Title: A Six Month Open Label Study of Amiloride Solution for Inhalation and Tobramycin Solution for Inhalation for the Eradication of Burkholderia Dolosa in Patients With Cystic Fibrosis
Brief Title: Amiloride Solution and Tobramycin Solution for Inhalation for the Eradication of Burkholderia Dolosa in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Dawn Ericson, MD, Children's Hospital, Boston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-06-0290
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Amiloride Solution for Inhalation — 4.5 mL, Amiloride Solution for Inhalation, Inhaled via Omron Ultrasonic Nebulizer, TID, 6 months

SUMMARY:
The purpose of this research study is to determine if multiple doses of two inhaled drugs will help Cystic Fibrosis patients whose lungs are infected with a bacteria called Burkholderia dolosa. The names of these drugs are tobramycin solution for inhalation and amiloride solution for inhalation. Currently, treating patients with Burkholderia dolosa infections is challenging because the bacteria is resistant to antibiotics. Therefore, researchers are looking for drugs which, when taken with an antibiotic, will help the antibiotic to work more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cystic Fibrosis
* Two positive cultures for Burkholderia dolosa lung infection

Exclusion Criteria:

* Positive pregnancy test or currently breast feeding (if applicable)
* Known sensitivity to Amiloride

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Eradication of Burkholderia dolosa. | 1 month, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Ericson, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital, Boston, Massachusetts, United States